CLINICAL TRIAL: NCT01199653
Title: Nonoperative Versus Operative Treatment of Midshaft Clavicle Fractures - A Randomized Controlled Trial
Brief Title: Study Comparing Plate Stabilization to Conservative Treatment in Midshaft Clavicle Fractures
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Kaisa Virtanen, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TYH6267; T102020Z12 (Other: Helsinki University Central Hospital)
Record Dates: First submitted 2010-09-10; First posted 2010-09-13 (Estimated); Last update posted 2010-09-13 (Estimated); Status verified 2010-09

CONDITIONS: Clavicle; Fracture
Keywords: clavicle fractures; midshaft; dislocated; operative treatment; conservative treatment; non-operative treatment; randomized controlled trial; bone plates
MeSH Terms: conditions — Fractures, Bone; Joint Dislocations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-operative treatment (Active Comparator): Non-operative (conservative) treatment of the clavicle fracture
  Interventions: Procedure: Non-operative treatment with arm immobilised to a sling
- Operative treatment (Active Comparator): Operative stabilization (i.e. ORIF) of the fracture with a plate and screws.
  Interventions: Procedure: Operative treatment

INTERVENTIONS:
Procedure: Operative treatment — Fracture stabilization with stainless steel reconstruction plate and screws. After the operation arm is immobilized to a sling for three weeks. Pendulum movements are allowed immediately.
  Arms: Operative treatment
Procedure: Non-operative treatment with arm immobilised to a sling — Arm is immobilised to a sling for three weeks. Pendulum movements are allowed immediately.
  Arms: Non-operative treatment

SUMMARY:
The purpose of this study is to find whether to operate or treat conservatively dislocated midshaft clavicle fractures.

DETAILED DESCRIPTION:
Midshaft clavicle fractures are common comprising 2% of all fractures and 35% to 45% of all shoulder girdle injuries in adults. Old-established treatment practices, based on no randomised controlled trials, are used for clavicle fractures. By tradition, midshaft clavicle fractures have been treated conservatively with arm immobilized to a sling for few weeks. The goal of treatment is to restore painless function of the upper extremity.

There have been some recommendations for operative treatment, such as skin compromising in fracture area, open fracture, floating shoulder, neurovascular symptoms in upper extremity, or multiple injuries. Recently, increasing interest has emerged in the surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* a completely displaced middle third clavicle fracture, no cortical contact between main fragments
* fresh fracture, treatment within seven days after injury
* age between 18 and 70 years
* provided informed consent

Exclusion Criteria:

* fracture was not dislocated
* multiple injured patient
* associated neurovascular injury, or suspicion of it
* reduced cooperation
* cancer or any severe illness impairing health
* pathological fracture
* treatment seven days after injury
* open fracture
* corticosteroid or immunosuppressive medication
* upper extremity fracture at same time
* an earlier clavicle or shoulder region fracture
* pregnancy
* lack of consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-08; Primary Completion 2007-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Shoulder function | Three months
  Shoulder Function is measured by Constant shoulder Score (CS) is a outcome measure for assessing the outcomes of the treatment of shoulder disorders.It inclues the pain score, functional assessment, range of motion and strength measures.
Shoulder function | One year
  Shoulder Function is measured by Constant shoulder Score (CS) is a outcome measure for assessing the outcomes of the treatment of shoulder disorders.It inclues the pain score, functional assessment, range of motion and strength measures.
Shoulder function | Two years
  Shoulder Function is measured by Constant shoulder Score (CS) is a outcome measure for assessing the outcomes of the treatment of shoulder disorders.It inclues the pain score, functional assessment, range of motion and strength measures.

SECONDARY OUTCOMES:
Disability of the Arm, Shoulder and Hand (DASH) | Three months
  The DASH is a self-report questionnaire designed to measure physical function and symptoms in people with any of several musculoskeletal disorders of the upper limb.
Pain at rest and activity | Three weeks
  Pain in measured with Visual Analogue Scale (VAS) which is a psychometric response scale. It is a measurement instrument for subjective characteristics that cannot be measured directly.
Fracture healing | Three months
  Fracture healing is examined from Xray.
Complications | Continous till two years
  Number of participants who are confronted complications such as nonunion, malunion, infection, hardware breakdown or hardware irritation.
Disability of the Arm, Shoulder and Hand (DASH) | One year
  The DASH is a self-report questionnaire designed to measure physical function and symptoms in people with any of several musculoskeletal disorders of the upper limb.
Disabilities of the Arm, Shoulder and Hand (DASH) | Two years
  The DASH is a self-report questionnaire designed to measure physical function and symptoms in people with any of several musculoskeletal disorders of the upper limb.
Pain at rest and activity | Six weeks
  Pain in measured with Visual Analogue Scale (VAS) which is a psychometric response scale. It is a measurement instrument for subjective characteristics that cannot be measured directly.
Pain at rest and at activity | Three months
  Pain in measured with Visual Analogue Scale (VAS) which is a psychometric response scale. It is a measurement instrument for subjective characteristics that cannot be measured directly
Pain at rest and at activity | One year
  Pain in measured with Visual Analogue Scale (VAS) which is a psychometric response scale. It is a measurement instrument for subjective characteristics that cannot be measured directly
Pain at rest and at activity | Two years
  Pain in measured with Visual Analogue Scale (VAS) which is a psychometric response scale. It is a measurement instrument for subjective characteristics that cannot be measured directly
Fracture healing | One year
  Fracture healing is examined from Xray.
Fracture healing | Two years
  Fracture healing is examined from Xray.

CONTACTS AND LOCATIONS:
Overall Officials: Kaisa J Virtanen, MD, Principal Investigator — Helsinki Uiversity Central Hospital; Ville Remes, MD PhD, Study Chair — Helsinki University Central Hospital; Jarkko Pajarinen, MD PhD, Study Chair — Helsinki University Central Hospital; Vesa Savolainen, MD PhD, Study Chair — Helsinki University Central Hospital; Jan-Magnus Björkenheim, MD PhD, Study Chair — Helsinki University Central Hospital; Mika P Paavola, MD PhD, Study Director — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Töölö Hospital, Helsinki, Uusimaa, Finland

REFERENCES:
- [Background] Canadian Orthopaedic Trauma Society. Nonoperative treatment compared with plate fixation of displaced midshaft clavicular fractures. A multicenter, randomized clinical trial. J Bone Joint Surg Am. 2007 Jan;89(1):1-10. doi: 10.2106/JBJS.F.00020. PMID 17200303
- [Background] Hill JM, McGuire MH, Crosby LA. Closed treatment of displaced middle-third fractures of the clavicle gives poor results. J Bone Joint Surg Br. 1997 Jul;79(4):537-9. doi: 10.1302/0301-620x.79b4.7529. PMID 9250733
- [Background] McKee MD, Seiler JG, Jupiter JB. The application of the limited contact dynamic compression plate in the upper extremity: an analysis of 114 consecutive cases. Injury. 1995 Dec;26(10):661-6. doi: 10.1016/0020-1383(95)00148-4. PMID 8745801
- [Background] NEER CS 2nd. Nonunion of the clavicle. J Am Med Assoc. 1960 Mar 5;172:1006-11. doi: 10.1001/jama.1960.03020100014003. No abstract available. PMID 14426324
- [Background] Nordqvist A, Petersson C. The incidence of fractures of the clavicle. Clin Orthop Relat Res. 1994 Mar;(300):127-32. PMID 8131324
- [Background] Nowak J, Holgersson M, Larsson S. Can we predict long-term sequelae after fractures of the clavicle based on initial findings? A prospective study with nine to ten years of follow-up. J Shoulder Elbow Surg. 2004 Sep-Oct;13(5):479-86. doi: 10.1016/j.jse.2004.01.026. PMID 15383801
- [Background] Nowak J, Mallmin H, Larsson S. The aetiology and epidemiology of clavicular fractures. A prospective study during a two-year period in Uppsala, Sweden. Injury. 2000 Jun;31(5):353-8. doi: 10.1016/s0020-1383(99)00312-5. PMID 10775691
- [Background] Poigenfurst J, Rappold G, Fischer W. Plating of fresh clavicular fractures: results of 122 operations. Injury. 1992;23(4):237-41. doi: 10.1016/s0020-1383(05)80006-3. PMID 1618563
- [Background] Zlowodzki M, Zelle BA, Cole PA, Jeray K, McKee MD; Evidence-Based Orthopaedic Trauma Working Group. Treatment of acute midshaft clavicle fractures: systematic review of 2144 fractures: on behalf of the Evidence-Based Orthopaedic Trauma Working Group. J Orthop Trauma. 2005 Aug;19(7):504-7. doi: 10.1097/01.bot.0000172287.44278.ef. PMID 16056089